CLINICAL TRIAL: NCT02035566
Title: Effectiveness of Telehome Monitoring on Quality of Life and Health Resources Utilization Among People With Chronic Disease Residing in Rural Maryland
Brief Title: Telehome Monitoring for Chronic Disease Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Claudia Baquet, Associate Dean and Professor Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00044150; RC2MD004800 (NIH)
Record Dates: First submitted 2013-01-16; First posted 2014-01-14 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Heart Failure; Pulmonary Disease, Chronic Obstructive; Hypertension; Diabetes Mellitus
Keywords: Minority Health; Health Status Disparities; Health Care Disparities; Rural Health; Telemedicine; Health Services Research; Social Determinants of Health; Ecological Theory of Health
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telehome Care Monitoring + Usual Care (Experimental)
  Interventions: Other: Telehome Care Monitoring
- Usual Care (No Intervention)

INTERVENTIONS:
Other: Telehome Care Monitoring — Telehome care monitoring over a 60-day period wherein patients transmit health measurements to their health care professional on a daily basis
  Arms: Telehome Care Monitoring + Usual Care

SUMMARY:
People living in rural areas are at increased risk for poor health outcomes due to: long distance to health care facilities, less available health care resources such as primary care and specialty services, transportation problems, higher elderly population, poverty, high uninsured rates and the lack of timely access to new technologies. Called Telehome Care (THC), in the form of equipment in the home, may provide an innovative and potentially cost-effective solution to enhancing chronic disease management services using technology and may influence the reduction in emergency department (ED) visits and hospitalizations in rural areas. However, telehealth research is still in its infancy, it is not well understood, and is often done without an overarching scientific framework. The provision of in home health monitoring and health education also may be a potential population based health research tool for chronically ill patients. Demonstration of the possible benefits, patient acceptance and satisfaction with THC requires a scientific approach as is used in this study.

DETAILED DESCRIPTION:
While the nation's overall health status has improved over the past decade, disparities persist among racial/ethnic minorities, low-income whites, the medically under-served, and rural residents. The disparities in disease morbidity and mortality are a compelling crisis and the elimination of such disparities is a national priority. With an aging population, the changing demographics are increasing the disease burden attributable to chronic diseases.

The broad goal of this project is to evaluate the potential value of using THC technology in chronically ill patients in rural Maryland, within the broad context of social determinants of health. This builds upon a completed pilot research study in Garrett County on a small scale THC program in rural Garrett County Maryland funded by the Maryland Cigarette Restitution Fund (CRF) supported Other Tobacco Related Diseases (OTRD grant) (CBaquet PI) in collaboration with the division of cardiology and department of family medicine. This research study will look at whether the THC equipment in the home for 60 days will make a difference in the health of the patients who get the unit in their home compared to the patients who will not receive the unit for 60 days. And we will look at whether this technology will support patient monitoring in the home. The use of the technology will be evaluated to determine whether patient monitoring using THC equipment will influence the hospitalization rates or emergency department visits for the patients. Evaluation of the influence of the THC equipment on medical resource utilization in rural and medically underserved communities will be studied.

Telehome care (THC) may provide augmentation to current face to face monitoring through home visits (usual method for Center for Medicaid and Medicare Services (CMS) billable home health services) of chronically ill patients and may provide an innovative and potentially cost-effective solution to improving patients' outcomes and health care resource utilization in rural areas. THC can support the coordination of care by assessing and monitoring patients in their homes and giving health care providers appropriate feedback to assure patient compliance with discharge instructions such as medication, home care and other aspects of recommended treatment regimens. Further, THC may improve service coordination at discharge and provide ongoing monitoring/engagement of patients, which is considered essential to prevent re-hospitalizations and emergency department visits. Demonstration of the potential benefits on care pathways, and patient and provider acceptance and satisfaction with the technology requires systematic larger scale and scientifically rigorous studies.

Purpose The project's broad goals are to evaluate the effects of telehome care (THC), a form of remote patient home monitoring,(within the broad context of social determinants of health) for chronic disease management among rural residing minority, low-income white, and medically underserved patients by: (a) providing an innovative telehome care (THC) capacity and infrastructure in two Maryland rural and medically underserved communities; and (b) using the THC infrastructure to generate scientifically rigorous and high quality evidence on whether the THC technology improves patient monitoring, influences clinical outcomes, and has an impact on medical resource utilization. [NOTE: THC uses telecommunication technologies to enable home health agency clinical staff at a rural home health agency to monitor their patients in the home.]

The major aim for this study are: 1) To evaluate the impact of the 60-day in home THC monitoring on medical resource utilization (emergency department visits; re-hospitalization rates) and Quality of Life related to the management of Metabolic Syndrome/Diabetes Mellitus (DM), Chronic Heart Failure (CHF), Hypertension (HTN), and Chronic Obstructive Pulmonary Disease (COPD) compared to those patients that receive only an educational pamphlet. Secondary aim hopes to support patient education to enhance acceptability, patient independence and satisfaction.

In this study, remote in-home patient monitoring using a THC system from VitelNet (telehealth equipment vendor) will provide patient monitoring remotely or non billable services for the experimental study arm for this project in addition to routine billable home health services. This project does not substitute billable in-home monitoring of patients which is a prerequisite for enrollment into this study(conventional home health services) but provides remote monitoring for the study arm in addition to conventional/billable services delivered.

Patients are randomized to either THC use for 60 days with 60, 90 day follow up or "usual care" with 60, 90 day follow up.

In addition, new knowledge will be generated by this study on methods for conduct of health disparities research and training of non-research clinical personnel who are community based in data collection and research ethics.

ELIGIBILITY:
Inclusion Criteria:

* Home bound at a home health agency (i.e., Garrett County Health Department Home Health Agency or Chesapeake-Potomac Home Health Agency)
* Clinical diagnosis of at least one of the following: chronic obstructive pulmonary disease, chronic heart failure, uncontrolled hypertension, diabetes mellitus and taking anti-hyperglycemic oral therapy
* Able to operate the telehome care system
* Agreeable to have the telehome care system installed at residence for 60 days
* Residing in an environment where care can be provided safely

Exclusion Criteria:

* Not eligible for home health care
* With a clinical diagnosis of a medical condition other than obstructive pulmonary disease, chronic heart failure, uncontrolled hypertension, diabetes mellitus and taking anti-hyperglycemic oral therapy
* Unable to follow instructions about or be able to operate the telehome care system
* Residing in an environment that is unsafe to provide home health care

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Self reported Quality of life | The Outcome Measure(s) are assessing a change from Baseline and 90-day post-baseline
  Assessing change from baseline to 90 day evaluated.
Number of emergency department visits | The Outcome Measure(s) are assessing a change from Baseline and 90-day post-baseline
  Assessing change from baseline to 90 day post baseline for:
  * exacerbation of a recent or remote diagnosis of chronic heart failure (post-baseline) requiring emergency department visit
  * exacerbation of chronic obstructive pulmonary disease (post-baseline) requiring emergency department visit
  * episodes of uncontrolled hypo/hyperglycemia (post-baseline) requiring emergency department visit
  * episodes of severe hypertension (post-baseline) requiring emergency department visit
Re-hospitalization | Assessing change from baseline and 90-day post-baseline
  Assessing change from baseline to 90 day post baseline for:
  * exacerbation of a recent or remote diagnosis of chronic heart failure (post-baseline) requiring hospital management
  * exacerbation of chronic obstructive pulmonary disease (post-baseline)requiring hospital management
  * episodes of uncontrolled hypo/hyperglycemia requiring emergency hospital management
  * episodes of severe hypertension requiring hospital management

SECONDARY OUTCOMES:
Number of contacts (visits or phone calls) with health care providers | Assessing change from baseline and 90-day post-baseline
Adequacy of hypertension control | Measures change from baseline and 90-day post-baseline
  Measures change from baseline to 90 day post baseline for:adequacy of blood pressure control (<140/90 mmHg)
Adequacy of diabetes control | Measures change from baseline and 90-day post-baseline
  adequacy of glycemic control of HbA1C of <7.5
Compliance with recommended (by discharging physician/primary health professional) drug therapy use for heart failure | Assessing change from baseline and 90-day post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Claudia R Baquet, MD MPH, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - Chesapeake-Potomac Home Health Agency, Hughesville, Maryland
  - Garrett County Health Department Home Health Agency, Oakland, Maryland